CLINICAL TRIAL: NCT05954910
Title: The Effectiveness and Safety of Polatuzumab in Real-World Clinical Practice Among Chinese Adult Patients With Diffuse Large B-Cell Lymphoma: A Prospective, Observational, Multicenter, Registry Study
Brief Title: A Study to Evaluate the Effectiveness and Safety of Polatuzumab in Real World Clinical Practice Among Adult Chinese Participants With Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML44616
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Unfit/frail participants with DLBCL who are untreated before the administration of polatuzumab and who have started receiving polatuzumab at physician's discretion in accordance with local clinical practice and/or labeling will be observed for safety and efficacy until death, withdrawal of consent, loss to follow-up or end of study whichever occurs first (up to approximately 3 years).
  Interventions: Drug: Polatuzumab Vedotin
- Cohort 2: Participants with DLBCL who can not be classified into unfit/frail but are untreated before the administration of polatuzumab and who have started receiving polatuzumab at physician's discretion in accordance with local clinical practice and/or labeling will be observed for safety and efficacy until death, withdrawal of consent, loss to follow-up or end of study whichever occurs first (up to approximately 3 years).
  Interventions: Drug: Polatuzumab Vedotin
- Cohort 3: Participants with relapsed or refractory (R/R) DLBCL who have started receiving polatuzumab at physician's discretion in accordance with local clinical practice and/or labeling will be observed for safety and efficacy until death, withdrawal of consent, loss to follow-up or end of study whichever occurs first (up to approximately 3 years).
  Interventions: Drug: Polatuzumab Vedotin

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Polatuzumab vedotin will be administered at the discretion of the physician per local clinical practice and local labeling.
  Other Names: POLIVY ®

SUMMARY:
The purpose of this study is to assess the progression free survival (PFS) in the real-world settings of polatuzumab among Chinese diffuse large B cell lymphoma (DLBCL) participants.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed as DLBCL
* Cohort 1: diagnosed as unfit/frail DLBCL. The unfit/frail is defined as aged 80 years or older, or younger than 80 years but with comorbidity and not tolerant to the standardized dose of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) therapy according to investigator's judgment
* Cohort 2: diagnosis as DLBCL but could not be classified into unfit/frail
* Cohort 3: relapse or refractory to previous treatment

Exclusion Criteria:

* Participant who currently participates in or with plan to participate in any interventional clinical trial
* Any other reason that, in the investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who will be treated with polatuzumab (known as being recommended and having the intention to be treated with polatuzumab at the time of signing informed consent) or have initiated polatuzumab treatment within three months prior to enrollment and after the indication approval will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Cohorts 1 and 2: Progression Free Survival at 24 months (PFS24) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | At 24 months
Cohort 3: PFS Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to end of study (EOS) (approximately 38 months)

SECONDARY OUTCOMES:
Cohort 3: PFS24 Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | At 24 months
Cohorts 1, 2 and 3: Time to Next Treatment (TTNT) | From the start of polatuzumab treatment to the initiation of next-line treatment (up to approximately 38 months)
Cohorts 1, 2 and 3: Complete Response Rate (CRR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to EOS (approximately 38 months)
Cohorts 1, 2 and 3: Overall Response Rate (ORR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to EOS (approximately 38 months)
Cohorts 1 and 2: Disease Control Rate (DCR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to EOS (approximately 38 months)
Cohorts 1, 2 and 3: Duration of Response (DoR) | From the date of the first occurrence of a documented CR or partial response (PR) to the date of progression, relapse, or death from any cause, whichever occurs first (up to approximately 38 months)
Cohorts 1 and 2: Disease Free Survival (DFS) | From the date of the first occurrence of a documented CR, to the date of relapse or death from any cause, whichever occurs first (up to approximately 38 months)
Cohorts 1 and 2: Event Free Survival (EFS) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | From the start of polatuzumab treatment to any treatment failure including disease progression, relapse, initiation of new antilymphoma therapy (NALT), or death from any cause, which occurs first (up to approximately 38 months)
Cohorts 1, 2 and 3: Overall Survival (OS) | From the start of polatuzumab treatment until the date of death from any cause (up to approximately 38 months)
Cohorts 1, 2 and 3: Number of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) | Up to EOS (approximately 38 months)
  AEs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (29):
- China (29):
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Hospital of Ministry of Health, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Xiangya Hospital of Centre-South University, Changsha
  - Third Xiangya Hospital of Central South University, Changsha
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu
  - Zhujiang Hospital, Southern Medical University, Guangzhou
  - Guizhou Cancer Hospital, Guiyang
  - Hainan Cancer Hospital, Haikou
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Jiangxi Cancer Hospital, Nanchang
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - The Affiliated Hospital Of Qingdao University, Qingdao
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Tongji Hospital of Tongji University, Shanghai
  - China Medical University (CMU) First Affiliated Hospital, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Province Cancer Hospital, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin Cancer Hospital, Tianjin
  - Xinjiang Medical University Cancer Hospital, Ürümqi
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Wuxi People's Hospital, Wuxi
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing